CLINICAL TRIAL: NCT05806866
Title: Progression in Cognition and Associated Activities of Daily Living (ADL) Impairment in Parkinson's Disease
Brief Title: Progression in Cognitive ADLs in Parkinson's Disease
Acronym: PRICOG-PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Technische Universität Dresden (Other); Luxembourg Institute of Health (Other Government); IB Hochschule für Gesundheit und Soziales (Unknown)
Responsible Party: Sponsor
Other Study IDs: 702/2022BO1
Record Dates: First submitted 2023-02-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Cognition; Actitvities of daily living function; Parkinson's disease dementia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid (CSF) samples will be collected in the morning, on an empty stomach. If patients do not agree for a lumbar puncture, fasting for blood sampling is not necessary for biomarker analysis.
  For patients with no CSF withdrawal about 40 ml venous blood will be collected for data analysis and storage of blood in the neurobank of the Hertie Institute for Clinical Brain Research (ethic proposal: 199/2011BO1). This amount does not represent any health hazard. Of those 10 ml of venous blood (1 Serum tube) will be used for study related analysis of neurofilament light chain. If the patient agrees for withdrawal of CSF additional 12,5 ml venous blood (2 serum tube, 1 glucose) will be taken for safety analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cognition scores, cognitive instrumental activities of daily living scores — A detailed neuropsychological test battery will be applied. The Functional Activitites Questionnaire (FAQ) subscores will be used to define cognitive and motor instrumental activities of daily living function

SUMMARY:
Mild cognitive impairment (PD-MCI) is one of the greatest risk factors for future Parkinson's disease dementia (PDD). A recent meta-analysis found that, on average, 31% of patients with PD-MCI converted to PDD within seven years; however, 24% of patients with PD-MCI reverted back to normal cognitive function. Consequently, the false positive rate for predicting PDD among patients with PD-MCI is high, and better predictive markers to define patients at high risk for PDD development are urgently needed. Therefore, a combination of different markers, including clinical, genetic, and other biomarker data, are proposed to increase ability to predict cognitive worsening and dementia. Based on data of the first follow-up of this cohort results indicated that presence of both mild cognitive instrumental activities of daily living (IADL) impairment and PD-MCI dramatically increases the risk for PDD (PubMed ID: 36240089). This study evaluates markers predicting cognitive and IADL long-term outcome in our sample. Additionally, focus of the study is the investigation whether ratings of patients or informants best predicted decline of cognitive impairment and/or everyday function. Clinical data along with other clinical marker and biomarker status will be investigated.

DETAILED DESCRIPTION:
Patients assessments: Most scales (except for Kölner Apraxie Test) were also included in the first follow-up of the sample. Total duration of scales and questionnaires is 4 hours (total time of mandatory in house assessments: 115 min).

Demographic and lifestyle data: Age, gender, education, occupation, family history of neurodegenerative diseases, smoking/drinking behavior, height & weight will be registered.

Activities of daily living assessment: The total and subscores of the Pfeffer Functional Activities Questionnaire (score range 0 to 30 higher values indicating more impairment) will be assessed. Additionally patients assessment includes the Parkinson's disease Activity of daily living scale (five level scale, higher values indicating more impairment).

Neuropsychological Assessment: History and self-awareness of cognitive deficits will be asked. Overall mean z-score (range -3.00 poor performance to +3.00 excellent performance) and cognitive domain score (mean z-score of tests assigned to one domain) will be quantitatively assessed using the Consortium to Establish a Registry for Alzheimer's Disease (CERAD-Plus) battery, three subtests of the Wechsler Intelligence Test for Adults (WIE), and one subtest of the Leistungsprüfsystem für 50- bis 90-Jährige (LPS 50+). The MMSE included in the CERAD-Plus, as well as the Montreal Cognitive Assessment (MoCA) will serve as global cognitive screening scales.

* Executive functions: Lexical and Phonemic Fluency (CERAD-Plus), Trail Making Test Part B (CERAD-Plus)
* Attention/working memory: Digit-Symbol Test (WIE), Letter-Number Sequencing (WIE)
* Language: Boston Naming Test (CERAD-Plus), Similarities (WIE)
* Memory: Word List Learning, Recall, and Discriminability (CERAD-Plus), Praxis Recall (CERAD-Plus)
* Visuospatial abilities: Praxis (CERAD-Plus), Fragmented Words (LPS-50+)

The Dementia Apraxia Test developed to assess limb and buccofacial apraxia in neurocognitive disorder patients with Alzheimer's disease and frontotemporal dementia will be additionally applied. For validation purpose, the Kölner Apraxie Screening will be included as well.

Clinical motor assessment: The Movement Disorder Society Unified Parkinson's disease rating scale (score 0 to 132) including the Hoehn and Yahr stage (score 0-5) will be applied. The Freezing of Gait Questionnaire (FOG) will be applied. Higher scale values indicated more severe impairment.

Additional non-motor assesssment: A comprehensive non-motor assessment will be applied including the Beck Depression Inventory II (BDI-II, score 0-63), the Beck Anxiety Scale (score 0-63), the Non-motor symptom Questionnaire (NMSQ, 0 to 30) and the Parkinson's disease Non-Motor Symptom Scale, subscales 1-5 (PD-NMS-S). In those scales higher values indicated more severe impairment.

Optional assessments:

* Blood withdrawal - 15 min
* Lumbar puncture - 30 min
* Ambulatory accelerometry device - 7 days

Caregiver assessments: To validate the patients' self-impression, caregiver questionnaires and interview scales will be applied, needing caregivers to be available for at least 38 minutes. Caregiver assessments will only be performed if the respective patient has agreed to the interview. The Bayer Activities of Daily Living Scale (1 point to 10 points with higher values indicating more impairment) answered by the caregiver and the Informant Questionnaire on Cognitive Decline in the Elderly (IQ-CODE, 26 points to 130 points, higher scores indicating more impaired performance) will be analysed.

ELIGIBILITY:
Between March 30th, 2014 and December 31th, 2017, a large cohort of 268 people with Parkinson's disease were recruited within the frame of the" Amyloid-Beta in cerebrospinal fluid as a risk factor for cognitive dysfunction in Parkinson's Disease" (ABC-PD) study. First follow-up was conducted between July 2018 and September 2020, including 182 (67.9%) patients. Those people with Parkinson's disease will be invited to participate in the proposed second follow-up assessment. If people with Parkinson's disease are not able to attend a clinical visit in-house, possibility of assessments at patients' homes shall be offered.

If people with Parkinson's disease or legal guardians give their consent a caregiver with regular contact to the patients will be ask to give information about patients instrumental activities of daily living, motor and non-motor status.

Inclusion Criteria:

* Participant in the " Amyloid-Beta in cerebrospinal fluid as a risk factor for cognitive dysfunction in Parkinson's Disease" (ABC-PD) study
* Diagnosis of Parkinson's disease according to the United Kingdom Brain Bank criteria.
* Ability to communicate well with the investigator, to understand and comply with the requirements of the study.
* Provide written informed consent to participate in the study and understand the right to withdraw consent at any time without prejudice to future medical care.
* If people with Parkinson's disease are not able to give consent for study participation (confirmed by an independent physician), study consent of a legal guardian is required.

Exclusion Criteria:

* Any disability that may prevent the subject from completing the informed consent form or other study requirements.
* Other neurodegenerative disease which renders the subject unable to communicate well with the investigator or to understand and comply with the requirements of the study.
* Participation in any clinical investigation of a new investigational compound or therapy within 4 weeks prior to baseline visit, and any other limitation of participation based on local regulations.
* Alcohol, medication, or drug dependency or abuse (except for nicotine).
* History of brain disease other than Parkinson's disease, e.g., head trauma, stroke, encephalitis.

Ages: 50 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants of the already recruited cross-sectional cohort will be asked to participate in the follow-up assessment. People with Parkinson's disease who did not agree to participate in a longitudinal study or who have asked not to be contacted after the first cross-sectional assessment will not be contacted again. A drop-out rate of 20% is expected for follow-up retention. Therefore, investigation of 145 people with Parkinson's disease will be primarily conducted between January 2023 and June 2024. During the executive project phase, around 7 to 9 patients will be assessed per month. People with Parkinson's disease will be contacted either via phone or in written form. Reasons for drop-outs will be registered for data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Parkinson's disease dementia (PDD) / Level II diagnosis of mild cognitive impairment in Parkinson's disease (PD-MCI) | 6-8 years
  Patients will be classified as PD-MCI according to Level-II Movement Disorder Society recommendations if cognitive impairment was present but did not significantly interfere with everyday function [PubMed ID: 21661055] according to a personalized interview. PDD was defined according to Movement Disorder Society Task Force criteria [PubMed ID: 18098298] if cognitive impairment was present and severe enough to impair activities of daily living function unrelated to motor or autonomic symptoms. Cognitive impairment will be defined according to Level-I (impairment of global cognition) for patients with minimal assessments, or Level-II (performance below 1.5 standard deviation of the population mean reported in the test manuals on at least two tests) for patients assessed using a full cognitive battery. Assessment include a detailed neuropsychological test battery (see below).

SECONDARY OUTCOMES:
Pfeffer Activities of daily living scale | 6-8 years
  Baseline/follow-up comparison of instrumental activities of daily living (IADL) function (patients' self-impression vs. informant-rating) primarily based on the motor, cognitive and total score of the Pfeffer Activities of daily living scale.
Follow-up score in global cognition | 6-8 years
  Overall mean z-score (range -3.00 poor performance to +3.00 excellent performance) of all tests assessed will be used to define global cognitive performance. For people with Parkinson's disease and incomplete neuropsychological test scores the MoCA will be used to define global cognitive performance.
Follow-up cognitive domain performance | 6-8 years
  Mean z-score of tests assigned to one cognitive domain will be used to define domain specific change in cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Inga Liepelt-Scarfone, PhD, Principal Investigator — Eberhard Karls Universität Tübingen
Locations (1):
- University hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol
Time Frame: During conduct and analysis
Access Criteria: Access will be granted upon reasonable request.

REFERENCES:
- [Background] Litvan I, Aarsland D, Adler CH, Goldman JG, Kulisevsky J, Mollenhauer B, Rodriguez-Oroz MC, Troster AI, Weintraub D. MDS Task Force on mild cognitive impairment in Parkinson's disease: critical review of PD-MCI. Mov Disord. 2011 Aug 15;26(10):1814-24. doi: 10.1002/mds.23823. Epub 2011 Jun 9. PMID 21661055
- [Background] Dubois B, Burn D, Goetz C, Aarsland D, Brown RG, Broe GA, Dickson D, Duyckaerts C, Cummings J, Gauthier S, Korczyn A, Lees A, Levy R, Litvan I, Mizuno Y, McKeith IG, Olanow CW, Poewe W, Sampaio C, Tolosa E, Emre M. Diagnostic procedures for Parkinson's disease dementia: recommendations from the movement disorder society task force. Mov Disord. 2007 Dec;22(16):2314-24. doi: 10.1002/mds.21844. PMID 18098298
- [Background] Becker S, Pauly C, Lawton M, Hipp G, Bowring F, Sulzer P, Hu M, Kruger R, Gasser T, Liepelt-Scarfone I. Quantifying activities of daily living impairment in Parkinson's disease using the Functional Activities Questionnaire. Neurol Sci. 2022 Feb;43(2):1047-1054. doi: 10.1007/s10072-021-05365-1. Epub 2021 Jun 10. PMID 34109514
- [Background] Becker S, Bode M, Brockmann K, Gasser T, Michaelis K, Solbrig S, Nuerk HC, Schulte C, Maetzler W, Zimmermann M, Berg D, Liepelt-Scarfone I. Cognitive-Driven Activities of Daily Living Impairment as a Predictor for Dementia in Parkinson Disease: A Longitudinal Cohort Study. Neurology. 2022 Dec 5;99(23):e2548-e2560. doi: 10.1212/WNL.0000000000201201. PMID 36240089

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT05806866/Prot_SAP_000.pdf